CLINICAL TRIAL: NCT01830257
Title: Phase 4 Study of MR and APDT Vaccine
Brief Title: Explore Active Surveillance Mode of the Community's Adverse Event Following Immunization(AEFI)
Acronym: AEFI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Beijing Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BJCDPC-7
Record Dates: First submitted 2013-03-31; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Adverse Reaction to Drug
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sending message (Experimental): The investigators would send the tip to the children's guardian
  Interventions: Other: sending message

INTERVENTIONS:
Other: sending message — Sending the suggestive short message

SUMMARY:
The investigators would remind the guardians of observation after immunization via sending short message and collect the information of AEFI by two ways, short message/telephone and website questionnaire.

DETAILED DESCRIPTION:
The investigators will compare the rate between active and inactive surveillance of AEFI

ELIGIBILITY:
Inclusion Criteria:

* According with the regular vaccination
* Immunization the acellular pertussis diphtheria tetanus vaccine and Measles and rubella combined vaccine

Exclusion Criteria:

* Disapproval the AEFI information

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Incidence about AEFI | 1.5years
  Incidence about AEFI comes from the rate between number of adverse event and the all quantity for immunization about MR and APDT

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoyun Wang, Doctor, Principal Investigator — Beijing Chaoyang District Centers for Disease Control and Prevention